CLINICAL TRIAL: NCT04483869
Title: Infrared Thermography and Apgar Score: Evaluation in Delivery Room for Term Newborn
Brief Title: Infrared Thermography and Apgar Score
Acronym: VIRGINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poissy-Saint Germain Hospital (Other)
Responsible Party: Principal Investigator, Mathilde Letouzey, MD, Principal investigator, Poissy-Saint Germain Hospital
Other Study IDs: 2020-A00265-34
Record Dates: First submitted 2020-07-09; First posted 2020-07-23 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Newborn, Transient
Keywords: thermography; apgar score
MeSH Terms: interventions — Thermography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thermography — thermographic image a 1, 3, 5 et 10 minutes of life

SUMMARY:
Background: The Apgar score assesses the newborn's adaptation in the first minutes of life. It is rated between 0 and 10 by the midwife, at 1-3-5 and 10 minutes of life. A low Apgar score at 5 minutes of life is associated with increased neonatal mortality and neurological impairment. However, this score has limitations and its measurement remains subjective: it does not guide resuscitation actions in the event of poor adaptation, significant inter-observer variability in scoring, variations according to the physiological maturation of the newborn, in particular according to gestational age.

Infrared thermography is a rapidly developing imaging technique based on the measurement of infrared radiation. It is an accurate, reliable and easy instrument of providing rapid non-contact, non-invasive and non-irradiating diagnosis. A recent 2018 study showed that the use of thermography would allow accurate and non-invasive monitoring of newborns in neonatal intensive care unit for early diagnosis of certain pathologies such as infection. During the transition, during the first minutes of life, the circulatory and respiratory systems of the newborn change. Vasodilatation occurs progressively in the central and peripheral areas. Thermoregulation is also a crucial stage of adaptation.

In view of this physiopathological knowledge, it seems interesting to correlate this adaptation , with the analysis of thermographic images. The principle of this technique is indeed based on the analysis of the heat emitted, and would thus make it possible to evaluate the blood perfusion of the newborn, and its evolution in the first minutes of life in an objective way. Our hypothesis is that a poor adaptation could be detected more efficiently on photographs taken at time T, contrary to the calculation of the Apgar score for which there are several limitations mentioned above.

Main objective of the study: To study the ability of the thermographic image to objectively evaluate the adaptation to ectopic life of newborns compared to existing evaluations (Apgar, pH, Lactates).

ELIGIBILITY:
Inclusion Criteria:

* term infants, gestational age ≥ 37 weeks of gestation
* cesarean delivery
* maternal age ≥ 18 years

Exclusion Criteria:

* parents refusal
* congenital anomalies

Max Age: 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term newborn, born after cesarean delivery, without congenital anomalies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
thermographic image | 1 minute of life
  Correlation between thermographic image and Apgar score
thermographic image | 5 minutes of life
  Correlation between thermographic image and Apgar score
thermographic image | 10 minutes of life
  Correlation between thermographic image and Apgar score

CONTACTS AND LOCATIONS:
Locations (1):
- Poissy Saint Germain Hospital, Poissy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Letouzey M, Diop S, Kengoum CEP, Rousseau A, Hot N, Francois J, Quibel T, Berveiller P, Boileau P, Jouen F, Trabelsi I, Bergounioux J. Newborn clinical condition assessment using infrared thermography: correlation with the Apgar score in a prospective cohort study. Front Pediatr. 2025 Dec 12;13:1636667. doi: 10.3389/fped.2025.1636667. eCollection 2025. PMID 41458084